CLINICAL TRIAL: NCT05997095
Title: Optimisation of Post-operative Electrical Muscle Stimulation (PoEMS) to Stimulate Muscle Protein Synthesis in Humans
Brief Title: Post-operative Electrical Muscle Stimulation to Stimulate Muscle Protein Synthesis in Humans
Acronym: PoEMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor of Translational Physiology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FMHS 261-0423
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Skeletal Muscle Atrophy
Keywords: Muscle; Protein Synthesis; Neuromuscular electrical stimulation; Muscle blood flow
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 30Hz (low-intensity) (Active Comparator): Volunteers receive 30 mins of neuromuscular electrical stimulation at 30Hz with a contraction pattern of 1 second "on" and 1 second "off"
  Interventions: Other: Neuromuscular electrical stimulation (NMES/0
- 100Hz (higher-intensity) (Experimental): Volunteers receive 30 mins of neuromuscular electrical stimulation at 100Hz with a contraction pattern of 1 second "on" and 1 second "off"
  Interventions: Other: Neuromuscular electrical stimulation (NMES/0
- 30Hz (low-intensity, 3:1) (Experimental): Volunteers receive 30 mins of neuromuscular electrical stimulation at 30Hz with a contraction pattern of 3 seconds "on" and 1 second "off"
  Interventions: Other: Neuromuscular electrical stimulation (NMES/0

INTERVENTIONS:
Other: Neuromuscular electrical stimulation (NMES/0 — NMES will be applied for 30 min and will be delivered using an approved, CE-marked device (Premier Combo Plus, Med-Fit Ltd, UK) using two large (7.5 × 13 cm) electrodes placed proximally and distally over the lateral quadriceps. The set protocols will be pre-programmed into to the device and the amplitude value will match the setting that was determined during a familiarisation visit

SUMMARY:
Skeletal muscle accounts for approximately 45-55% of total body mass in healthy adults and plays a pivotal role in whole-body metabolic health, locomotion and physical independence. Undesirable loss of skeletal muscle mass (atrophy) is, however, a common feature of many communicable and non-communicable diseases including ageing, bed-rest/immobilisation, cancer and physical inactivity. As such, the design of optimal strategies (e.g., different types of exercise) to "offset" these detrimental losses of muscle is a focus for both researchers and clinicians.

One situation where losses of muscle mass occur very quickly (i.e., within a few days) is after surgery. However, at this time, most people (especially if they have had major abdominal or lower-limb surgery) are not able to perform exercise and as such a different strategy to maintain muscle mass needs to be found. It has been shown that electrical stimulation of the leg muscles can maintain muscle mass and function in patients after surgery. It is not however yet known, what the optimal electrical stimulation regime is to preserve muscle mass during situations of disuse.

This study aims to examine the impact of three different electrical stimulation protocols on muscle building processes in individuals age-matched to those most commonly presenting for major abdominal surgery. This information will then be used in a clinical trial of surgical patients to see if it can preserve their muscle mass and function in the post-operative period.

DETAILED DESCRIPTION:
The contraction of skeletal muscles depends on the regulation of the nervous system and the coordination of neuromuscular function. The smallest motor nervous system associated with muscle contraction is the motor unit (MU), which consists of an efferent motor neuron and all of the muscle fibres it innervates. Muscle tissue also undergoes adaptive alternations in response to external stimuli, such as the gradual decline in muscle mass and strength during ageing, and atrophy following muscle disuse. A number of studies have demonstrated that different types of voluntary movements, such as resistance exercise training (RET), can prevent or attenuate such alternations to a certain extent via increases in muscle protein synthesis (MPS).

However, certain situations such as post-operative bed rest render RET interventions an unachievable option. Neuromuscular electrical stimulation (NMES) can be applied as a surrogate; acting to evoke involuntary contraction of the target muscles via electrical current applied to the muscle belly. Although NMES stimulation has been widely tested in the intensive care environment, results have shown variable efficacy- perhaps due to the multi-organ failure and associated catabolic systemic environment encountered by the majority of these patients.

It has recently shown that in post-operative abdominal surgery patients, 5-days of NMES, performed at frequency of 30 Hz in a 1 second "on", 1 second "off" contraction pattern, can mitigate losses in muscle mass and function. However, this study 'borrowed' a protocol from previous intensive care literature, and as such may not be optimal with regards to frequency or contraction pattern. Given that this protocol was highly tolerated by patients in a previous study (i.e., based on 30 min of daily NMES, patients in this study said they would tolerate it for 45 to 240 (mean 90) min), it is plausible that higher frequency NMES (~100 Hz), enabling greater force production may be both viable and result in further mitigation of muscle mass and function losses. It has also been demonstrated that the time muscle is under loaded tension during RET may be an important modulator of MPS and subsequent gains in muscle mass. Therefore, increasing the contraction relative to relaxation time during NMES (e.g., 3 seconds on, 1 second off) may be another feasible and perhaps more beneficial strategy to reduce muscle mass losses in populations where an increase in frequency may not be possible or tolerable.

Knowing that muscle maintenance is based on a dynamic equilibrium between MPS and muscle protein breakdown, the impact of different NMES protocols on MPS, associated cell signalling, and nutrient delivery pathways needs to be explored so that an optimal intervention can be tested in clinical settings associated with disuse atrophy. To date, no previous studies have compared differing frequencies of NMES on the muscle metabolic responses in older adults, nor the effect of differing NMES-induced contraction patterns.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-85 y
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* BMI <18.5 or >35kg/m2
* Participation in any regular, structured RET within the past 6 months
* Musculoskeletal disorders
* Severe respiratory disease:
* COPD
* Pulmonary hypertension
* Neurological disorders:
* Cerebrovascular disease (cerebral haemorrhage; cerebral ischemic stroke)
* Intracranial space-occupying lesion
* Epilepsy
* Metabolic disease:
* Hyper and hypo parathyroidism
* Untreated hyper and hypothyroidism
* Cushing's disease
* Type 1 or 2 diabetes
* Active cardiovascular problems:
* Uncontrolled hypertension (BP>160/100mmHg)
* Recent cardiac event
* Heart failure (Class III/IV)
* Arrhythmia
* Angina
* Blood clotting disorders
* Active inflammatory bowel or renal disease
* Recent malignancy (in previous 3 years)
* Recent steroid treatment within 6 months or hormone replacement therapy
* Family history of early (<55yrs) death from cardiovascular disease
* Known sensitivity to Sonovue

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Protein Synthesis | 4 hours
  A primed continuous infusion of a stable isotope tracer (1,2 13C2] leucine) will be initiated (Prime: 0.7 mg/kg; Constant: 1.0 mg/kg/h) at time 0h. After 60 min of stable isotope infusion, a single muscle biopsy will be taken from one leg. Another biopsy from the same leg will be taken 120 min later, and a third 240 min after the second to provide rates of muscle protein synthesis in the rested condition and in response to NMES, respectively. The fractional synthetic rate (FSR) of the myofibrillar fraction was calculated from the incorporation of [1,2 13C2] leucine, using venous plasma labelling between muscle biopsies to represent the immediate precursor for protein synthesis. This will give a rate (%/hour) of muscle protein synthesis.

SECONDARY OUTCOMES:
Skeletal Muscle Anabolic Signalling | 4 hours
  Total and phosphorylation of established anabolic proteins in human skeletal muscle will be quantified via Western Blotting.
Skeletal Muscle Blood Flow | Baseline and 30 minutes post neuromuscular stimulation
  Contrast enhanced ultrasound (CEUS) measurements will be made 60 min before the NMES and 30 min after. To achieve this, a custom-made probe holder will be placed on the leg to be stimulated at the start of the study. For each measurement, Sonovue will be infused at 2ml/min for 1 minute and then 1ml/min for 30 sec to achieve systemic steady state, with a continued infusion at 1ml/min for the duration of the measurements. Each measurement will include three, 30-second capture-flash cycles which will form a Sonovue replenishment curve for the portion of vastus lateralis muscle (VL) under the probe. blood flow will be calculated by measuring the reperfusion rate of the microbubbles in the muscle microvasculature following destruction with a high mechanical index flash, given the infusion of contrast is continuous.

OTHER OUTCOMES:
Perceived discomfort of Neuromuscular Electrical stimulation | Immediately post neuromuscular stimulation
  At the end of the NMES, participants will be asked to rate the perceived discomfort on a Likert scale of 1-10 and respond to the question of "that stimulation was 30-minutes, how much longer would you have been willing to have stimulation for if you were in bed recovering from an injury or illness i.e., it was not interfering with your ability to perform other activities?"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy EJ, Hatt J, Doleman B, Smart TF, Piasecki M, Lund JN, Phillips BE. Post-operative electrical muscle stimulation attenuates loss of muscle mass and function following major abdominal surgery in older adults: a split body randomised control trial. Age Ageing. 2022 Oct 6;51(10):afac234. doi: 10.1093/ageing/afac234. PMID 36315433
- [Background] Hardy EJO, Inns TB, Hatt J, Doleman B, Bass JJ, Atherton PJ, Lund JN, Phillips BE. The time course of disuse muscle atrophy of the lower limb in health and disease. J Cachexia Sarcopenia Muscle. 2022 Dec;13(6):2616-2629. doi: 10.1002/jcsm.13067. Epub 2022 Sep 14. PMID 36104842
- [Background] Wall BT, Dirks ML, Verdijk LB, Snijders T, Hansen D, Vranckx P, Burd NA, Dendale P, van Loon LJ. Neuromuscular electrical stimulation increases muscle protein synthesis in elderly type 2 diabetic men. Am J Physiol Endocrinol Metab. 2012 Sep 1;303(5):E614-23. doi: 10.1152/ajpendo.00138.2012. Epub 2012 Jun 26. PMID 22739107
- [Background] Mancinelli R, Toniolo L, Di Filippo ES, Doria C, Marrone M, Maroni CR, Verratti V, Bondi D, Maccatrozzo L, Pietrangelo T, Fulle S. Neuromuscular Electrical Stimulation Induces Skeletal Muscle Fiber Remodeling and Specific Gene Expression Profile in Healthy Elderly. Front Physiol. 2019 Nov 27;10:1459. doi: 10.3389/fphys.2019.01459. eCollection 2019. PMID 31827446
- [Background] Burd NA, Andrews RJ, West DW, Little JP, Cochran AJ, Hector AJ, Cashaback JG, Gibala MJ, Potvin JR, Baker SK, Phillips SM. Muscle time under tension during resistance exercise stimulates differential muscle protein sub-fractional synthetic responses in men. J Physiol. 2012 Jan 15;590(2):351-62. doi: 10.1113/jphysiol.2011.221200. Epub 2011 Nov 21. PMID 22106173